CLINICAL TRIAL: NCT00105638
Title: A Telehealth Education Program for Caregivers of Veterans With Dementia
Brief Title: Telehealth Education Program for Caregivers of Veterans With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IIR 03-076
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-11

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Intervention studies; Health Care Costs; Telephone; Caregivers
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: educational program, by telephone

INTERVENTIONS:
Behavioral: educational program, by telephone

SUMMARY:
This study was designed to evaluate the impact of a Telehealth Education Program (TEP) on outpatient veterans with moderate to severe dementia and their spouse caregivers. The TEP is a program of education, coping skills, problem solving and support presented to caregivers of veterans with dementia by teleconference in 10 weekly, one-hour sessions. The TEP was based on a stress and coping model aimed to enhance the knowledge, skills and feelings of support of the caregivers who participated.

DETAILED DESCRIPTION:
Background:

This study was designed to evaluate the impact of a Telehealth Education Program (TEP) on outpatient veterans with moderate to severe dementia and their spouse caregivers. The TEP is a program of education, coping skills, problem solving and support presented to caregivers of veterans with dementia by teleconference in 10 weekly, one-hour sessions. The TEP was based on a stress and coping model aimed to enhance the knowledge, skills and feelings of support of the caregivers who participated.

Objectives:

The objectives of this study were to: 1) evaluate the impact of TEP on outpatient veterans with dementia; and 2) to help spousal caregivers gain the knowledge and skills necessary to provide the highest quality of care possible for their spouse in order to prevent unnecessary healthcare utilization and premature institutionalization. In addition, a second objective was to develop a TEP training manual for VA clinical staff and a TEP workbook for family members.

Methods:

This study employed a 2x3x2x4 randomized control group design. The design had two levels of intervention, TEP verus usual care(UC), three times of measurement (baseline, 3 months and 12 months), two sites of educational group intervention, (Albany VAMC and Buffalo VAMC) and four leaders (two nestled at each of the two sites). Veterans were included into the study if: 1) they were community dwelling; 2) had been diagnosed with Alzheimer's disease, or a related dementing disorder, and 3) scored three or higher on the Global Deterioration Scale. Caregivers were included if they: 1) were the primary care providers for the veterans, 2) had cohabitated with the veteran for more than one year, 3) reported at least a moderate level of strain, (score a seven or higher on the Caregiver Strain Index), and (4) had not participated in any other individual or group intervention program designed to support caregivers of demented persons.

There were ten TEP caregiver groups that received the educational program in one-hour sessions for 10 weeks. Demographic data were collected on the veterans and caregivers at baseline. Psychosocial outcome data were collected within two weeks prior to the intervention(baseline) and then again at three and twelve months. These were collected to evaluate whether TEP veterans would experience a reduction in behavioral problems, agitation and symptoms of depression and whether caregivers would experience a significant increase in dementia management skills, as well as, a perceived ability to care for their spouse. Outcome variables were analyzed using mixed effect regression models. Healthcare cost and utilization data were extracted from the VISTA databases and included outpatient, inpatient and nursing home data within the VA.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

* spouse of veteran
* clinical diagnosis of dementia/Alzheimers
* verbal approval from primary care provider
* living with partner

Exclusion Criteria:

* not spouse of veteran
* no clinical diagnosis of dementia
* no verbal approval from PCP
* not living with partner

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Reduction in veteran agitation and symptoms of depression; increase in caregiver management skills

SECONDARY OUTCOMES:
Veterans will experience fewer hospitalizations and nursing home admissions

CONTACTS AND LOCATIONS:
Overall Officials: Mollie Shulan, MD, Principal Investigator — Albany VA Medical Center Samuel S. Stratton, Albany, NY
Locations (2):
- United States (2):
  - Albany VA Medical Center Samuel S. Stratton, Albany, NY, Albany, New York
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York

REFERENCES:
- [Result] Wray LO, Shulan MD, Toseland RW, Freeman KE, Vasquez BE, Gao J. The effect of telephone support groups on costs of care for veterans with dementia. Gerontologist. 2010 Oct;50(5):623-31. doi: 10.1093/geront/gnq040. Epub 2010 May 27. PMID 20507926